CLINICAL TRIAL: NCT03250611
Title: Occipito-Cervical Stabilization Using Occipital Condyle as a Cranial Anchor
Brief Title: Occipito-Cervical Stabilization Using Occipital Condyle Screw
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Muhammad Almessry, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OC.Screw
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Cervical Instabilities Spine
Keywords: Occipital condyle; Occipital condyle screw

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Occipito-Cervical Instability (Experimental): Stabilization of the occipito-cervical junction by Occipital Condyle Screw (OCS) as a sole cranial anchor, with posterior bone graft.
  Interventions: Procedure: Occipital Condyle Screw

INTERVENTIONS:
Procedure: Occipital Condyle Screw — Occipito-Cervical Screw-Rod Fixation Technique

SUMMARY:
The Occipito-Cervical (OC) junction is the most cephalad portion of the spinal axis, with anatomical osseous complex that allows significant mobility while maintaining biomechanical stability. OC instability is a rare disorder with potentially life-threatening consequences. Instability may manifest as disabling pain, cranial nerve dysfunction, paralysis, or even sudden death. The most common acute presentation is secondary to major trauma. Other pathologic processes that may lead to chronic instability include rheumatoid arthritis, infections, tumors, and even congenital malformations; OC fusion in aforementioned cases each according is then indicated.

Stabilization of the OC junction remains a challenge, owing to the regional anatomy and poor occipital bone purchase. OC stabilization techniques have undergone continuous refinement. Early techniques involving simple posterior only bone grafts demonstrated a high rate of failure and have largely been replaced by rigid posterior fixation systems using rods/screws or plates, providing superior biomechanical stability and higher rates of fusion. One of the very modern modalities of fixation methods is the Occipital Condyle Screw (OCS) as a sole cranial anchor; believing that decreasing the length of lever arm of the construct, increasing the length of the screw purchase, and decreasing stresses addressed on the rod with no need to excessively bend it for the occipital slope may enhance the construct rigidity, and leaving a greater clear metal-free area of the occiput for graft contact may have a real potential benefits in fusion rates.

DETAILED DESCRIPTION:
Clinical Evaluation: of patients with 1- Visual Analogue Scale (VAS), 2- Neck Disability Index (NDI), 3- Modified Japanese Orthopaedic Association Cervical Myelopathy Score (mJOA.CMS), 4- American Spinal Injury Association Score (ASIAs). Immediate preoperative functional scoring, and 6 weeks, 3 months, 6 months, and 1 year postoperative.

Surgical Technique: The patient is handled in prone position after successful general anaesthesia with supported head to ensure that the Occipito-Cervical junction maintains in neutral position. The Occipito-Cervical junction is then exposed through a traditional midline longitudinal posterior skin incision extends from the external occipital protuberance to the C3-C4 level. The nuchal ligament is divided in the midline, and the occipital and cervical musculature is dissected subperiosteally. The suboccipital and cervical paraspinous muscles are retracted laterally to expose the underlying bony architecture. The posterior arch of C1 is exposed and the dissection is continued laterally in a subperiosteal manner to identify the horizontal segment of the vertebral arteries (VAs) which is enveloped in a dense venous plexus. The atlanto-occipital joint capsule is to be approx. 3 mm. Cranial to the superior margin of tht VA. Attention is then focused on the foramen magnum. Using curettes, the atlanto-occipital membrane is gently dissected from the foramen magnum laterally until the medial aspect of the occipital condyle is reached. At this point, the dissection continues laterally, maintaining bone contact to prevent injury to the horizontal segment of the VA along the condylar fossa, until the posterior condylar foramen and emissary vein are identified. The condylar foramen and vein represent the lateral extent of the dissection. At this stage, the operative field is prepared for instrumentation. Inserting the cervical screws first provides useful information about the axial location of the occipital condyles. The condylar entry point (CEP) is defined using a combination of radiographic and anatomic landmarks. The CEP is located (4 to 5 mm) lateral to the posteromedial edge of the condyle, and (2 mm) above the atlanto-occipital joint line. Pilot hole is then made at the entry point using an awl with slight cranial angulation to avoid injury to the horizontal segment of the VA. The pilot hole is then drilled under image-guidance in a convergent trajectory with (12 to 22 degrees) of medial angulation and (5 degrees) cranial angulation in the sagittal plane with the tip of the drill directed toward the basion, advancing slowly until the anterior cortical edge of the condyle is breached. The hole is tapped, and a (3.5 mm) polyaxial screw of an appropriate length (30 to 34 mm) is inserted bicortically into the occipital condyle. Approximately (12 mm) portion of the screw remains superficial to the posterior cortex of the condyle, allowing the polyaxial portion of the screw to lie above the posterior arch of C1, minimizing any chance of irritation of the VA by the rods.

Radiological Evaluation: 1- Preoperative: Plain X-ray (PXR) Antero-posterior (AP) and Lateral (Lat.) views to study the upper cervical instability indices and measurements, Multi-Slice Computed Tomography (MSCT) to study the boney Occipito-Cervical architecture for any fractures or anomalies, CT Angiography (CTA) to study the vertebral artery for anomaly especially in the horizontal segment of the VA, and Magnetic Resonance Imaging (MRI) to study the spinal cord for any compression signs. 2- Postoperative: Immediate (PXR) AP. and Lat. views for overall global assessment of the reduction and the construct installation. Then at 3 months, 6 months, and 1 year after surgery with flexion extension lateral view bending stress films for assessment of stability. Immediate (MSCT) to study the crucial screws placement estate for any breaches or successfulness, and after 1year for assessment of the fusion rate achieved.

Serial Follow-Up: after 6 weeks for clinical evaluation and functional scoring. At 3 and 6 months for radiological evaluation of stability, clinical evaluation and functional re-scoring. At 1 year for evaluation of fusion rate, clinical evaluation and over all resultant functional scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients with occipito-cervical instability of any cause, indicated for occipito-cervical fusion

Exclusion Criteria:

* Fractured occipital condyle
* Congenital malformation of occipital condyle
* Congenital anomaly of the horizontal segment of the vertebral artery

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
CT based classification for assessment of biological graft fusion | At 6 months postoperative
  A new assessment method of bony union using high-speed spiral CT imaging is proposed which reflects the gradually increasing biological stability of the construct. Grade I (complete fusion) implies cortical union of the allograft and central trabecular continuity. Grade II (partial fusion) implies cortical union of the structural allograft with partial trabecular incorporation. Grade III (unipolar pseudarthrosis) denotes superior or inferior cortical non-union of the central allograft with partial trabecular discontinuity centrally and Grade IV (bipolar pseudarthrosis) suggests both superior and inferior cortical non-union with a complete lack of central trabecular continuity.

SECONDARY OUTCOMES:
Visual Analogue Scale for Pain (VAS Pain) | Baseline measure, then at 2 weeks, 3 months and 6 months postoperative
  Operationally a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.
Neck Disability Index (NDI) | Baseline measure, then at 2 weeks, 3 months and 6 months postoperative
  Each of 10 items, which are 1. Pain intensity 2. Personal care 3. Lifting 4. Reading 5. Headaches 6. Concentration 7. Work 8. Driving 9. Sleeping 10. Recreation, is scored from 0 - 5. The maximum score is therefore 50. The obtained score can be multiplied by 2 to produce a percentage score. Occasionally, a respondent will not complete one question or another. The average of all other items is then added to the completed items.
  The original report provided scoring intervals for interpretation, as follows: 0 - 4 = no disability, 5 - 14 = mild, 15 - 24 = moderate, 25 - 34 = severe, and above 34 = complete.
American Spinal Injury Association Score (ASIAs) | Baseline and 3 months postoperative
  A score developed by the American Spinal Injury Association for essential minimal elements of neurologic assessment for all patients with a spinal injury.
  (A). Complete loss of motor and sensory function below the level of injury, including the anal saddle shaped area.
  (B). Spared all/some sensory function below the level of injury, including the anal saddle shaped area.
  (C). Spared all/some motor function below the level of injury, but cannot move against gravity.
  (D). Spared all/some motor function below the level of injury, with ability to move against gravity.
  (E). Neurologically free.
Modified Japanese Orthopaedic Association Cervical Spondylotic Myelopathy Score (mJOA.CSM) | Baseline and 3 months postoperative
  Motor dysfunction Upper extremities
  0. Doesn't move hands
  1. Doesn't eat with a spoon, moves hands
  2. Doesn't button shirt, eats with a spoon
  3. Buttons shirt with great difficulty
  4. Buttons shirt with slight difficulty
  5. No dysfunction
  Motor dysfunction Lower extremities
  0. Complete loss motor & sensory
  1. Sensory preservation, doesn't move legs
  2. Moves legs, doesn't walk
  3. Walks on flat floor with walking aid
  4. Walks up or downstairs w/aid of a handrail
  5. Moderate-to-significant lack of stability, walks up or downstairs without handrail
  6. Mild lack of stability, walks unaided with smooth reciprocation
  7. No dysfunction
  Sensory dysfunction Upper extremities
  0. Complete loss of hand sensation
  1. Severe sensory loss or pain
  2. Mild sensory loss
  3. No sensory loss
  Sphincter dysfunction
  0. Unable to micturate voluntarily
  1. Marked difficulty in micturition
  2. Mild-to-moderate difficulty in micturition
  3. Normal micturition

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed El-Meshtawy, MD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uribe JS, Ramos E, Vale F. Feasibility of occipital condyle screw placement for occipitocervical fixation: a cadaveric study and description of a novel technique. J Spinal Disord Tech. 2008 Dec;21(8):540-6. doi: 10.1097/BSD.0b013e31816d655e. PMID 19057245
- [Background] Uribe JS, Ramos E, Youssef AS, Levine N, Turner AW, Johnson WM, Vale FL. Craniocervical fixation with occipital condyle screws: biomechanical analysis of a novel technique. Spine (Phila Pa 1976). 2010 Apr 20;35(9):931-8. doi: 10.1097/BRS.0b013e3181c16f9a. PMID 20375778
- [Background] Uribe JS, Ramos E, Baaj A, Youssef AS, Vale FL. Occipital cervical stabilization using occipital condyles for cranial fixation: technical case report. Neurosurgery. 2009 Dec;65(6):E1216-7; discussion E1217. doi: 10.1227/01.NEU.0000349207.98394.FA. PMID 19934947
- [Background] La Marca F, Zubay G, Morrison T, Karahalios D. Cadaveric study for placement of occipital condyle screws: technique and effects on surrounding anatomic structures. J Neurosurg Spine. 2008 Oct;9(4):347-53. doi: 10.3171/SPI.2008.9.10.347. PMID 18939920
- [Background] Ahmadian A, Dakwar E, Vale FL, Uribe JS. Occipitocervical fusion via occipital condylar fixation: a clinical case series. J Spinal Disord Tech. 2014 Jun;27(4):232-6. doi: 10.1097/BSD.0b013e31825bfeea. PMID 24866907
- [Background] Tan GH, Goss BG, Thorpe PJ, Williams RP. CT-based classification of long spinal allograft fusion. Eur Spine J. 2007 Nov;16(11):1875-81. doi: 10.1007/s00586-007-0376-0. Epub 2007 May 12. PMID 17497188